CLINICAL TRIAL: NCT05396534
Title: Personalized Persistent Atrial Fibrillation Ablation: The PeAF-BY-LAWT Trial
Acronym: PeAF-by-LAWT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Medico Teknon (Other)
Responsible Party: Principal Investigator, Antonio Berruezo, MD, PhD, Head of Arrhythmia Department, Centro Medico Teknon
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PeAF-by-LAWT
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Persistent Atrial Fibrillation; Persistent Atrial Fibrillation Longstanding
Keywords: Atrial Fibrillation; Catheter Ablation; Multidetector Computed Tomography; Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Two-arm, single-blind, single-center, randomized controlled trial
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- byLAWT arm (Experimental): Personalized protocol that uses a contact-force catheter, a multichannel radiofrequency generator, and integrated MDCT-derived Left Atrial Wall Thickness (LAWT) information to adapt the ablation index target to the subjacent LAWT.
  Interventions: Procedure: Atrial Fibrillation transcatheter ablation
- CLOSE arm (Active Comparator): In the CLOSE arm, the use of MDCT-derived LAWT information will not be available for the operator. We uses a contact-force catheter. Ablation will be performed according to the CLOSE study settings: Power-controlled mode (without ramping) with 25 to 35 W (irrigation flow 30 ml/min). RF will be delivered until an AI of 400 at the posterior wall/roof an 550 at the anterior wall are reached.
  Interventions: Procedure: Atrial Fibrillation transcatheter ablation

INTERVENTIONS:
Procedure: Atrial Fibrillation transcatheter ablation — We perform pulmonary veins isolation that remains remains the cornerstone of all catheter-based treatment strategies in atrial fibrillation

SUMMARY:
The investigators hypothesized that PeAF-by-LAWT, a personalized protocol that uses a contact-force catheter, a multichannel radiofrequency (RF) generator, and integrated LAWT information to adapt the ablation index (AI) target to the subjacent LAWT, is safe, while showing at least the same efficacy and better efficiency than the CLOSE protocol for persistent AF ablation.

DETAILED DESCRIPTION:
Pulmonary vein isolation (PVI) remains the cornerstone of all catheter-based treatment strategies in atrial fibrillation (AF). Currently, PVI is recommended (class IA indication) after one failed or intolerant class I or III antiarrhythmic drug (AAD) to improve symptoms, either in paroxysmal (PaAF) or persistent AF (PeAF). However, PVI can be also considered as first-line treatment to achieve rhythm control, particularly in cases when tachycardia-induced cardiomyopathy is suspected, a circumstance likely more related to a higher AF burden or PeAF.

PVI has been proven to be effective in treating PeAF, although long-term ablation outcomes have been significantly less satisfactory than in PaAF. In a recent metaanalysis, PVI in PeAF achieved an arrhythmia-free survival at 12 months of 66.7%, with > 80% of the patients off AAD. Other ablation strategies combining PVI plus additional substrate ablation (linear ablation and/or complex fractionated atrial electrogram ablation) have been unable to demonstrate better outcomes than PVI-alone.

On the other hand, recent advances both in technology and ablation protocols have resulted in greatly improved outcomes after PVI. The introduction of contact force-sensing catheters, novel estimates of lesion size [ablation index (AI) or lesion size index, and the fact of ensuring lesion contiguity (≤ 6 mm inter-lesion distance) have markedly improved arrhythmia-free survival after PVI, particularly in PaAF.

The CLOSE clinical study analyzed the utility of ablation index (AI), a novel formula developed to assess real-time effect of RF delivery and improve the rates of PVI, with 91.3% of the patients free from AF/AT/atrial flutter (AFL) at 12 months follow-up. The CLOSE protocol targeted an interlesion distance (ILD) of 6 mm and AI ≥ 400 at the posterior wall and ≥550 at the anterior wall. Recently, Hussein et al. demonstrated that the use of AI-guided PVI alone performed with radiofrequency energy in a point-by-point wide area circumferential ablation (WACA) pattern according to CLOSE protocol achieves good clinical outcomes in persistent AF patients at 12 months follow-up. Finally, a more recent, personalized PVI strategy, aiming for contiguous lesions with AI titration according to the local left atrial wall thickness (LAWT) as per multidetector cardiac tomography (MDCT), has demonstrated to achieve an arrhythmia-free survival > 95% at 12 months in PaAF.

Up to date, there are no randomized studies for persistent AF ablation comparing the outcomes of PVI-alone procedures performed with a personalized ablation protocol that uses the information of left atrial wall thickness (LAWT), compared with the CLOSE protocol.

The investigators hypothesized that PeAF-by-LAWT, a personalized protocol that uses a contact-force catheter, a multichannel radiofrequency (RF) generator, and integrated LAWT information to adapt the ablation index (AI) target to the subjacent LAWT, is safe, while showing at least the same efficacy and better efficiency than the CLOSE protocol for persistent AF ablation.

This is a two-arm, single-blind, single-center, randomized controlled trial. The study will be conducted in a tertiary hospital with an electrophysiology team of qualified investigators with proven experience in performing atrial fibrillation ablation.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Indication for persistent atrial fibrillation ablation.
* Signed informed consent

Exclusion Criteria:

* Age < 18 years.
* Pregnancy.
* Previous AF redo procedure.
* Impossibility to perform a pre-procedural CT scan.
* Concomitant investigation treatments.
* Medical, geographical and social factors that make study participation impractical, and inability to give written informed consent. Patient's refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Arrhythmia-free survival | After the 3-month 'blanking period' for 12 month
  The efficacy primary endpoint will be survival free of any atrial arrhythmia at12-month follow-up visits. From this endpoint, important definitions must be taken into account: AF clinical recurrence will be considered only after the 3-month 'blanking period'.

SECONDARY OUTCOMES:
Procedure time | intraprocedural outcome
  Reduction of procedure time in the byLAWT arm
Radiofrequency time | intraprocedural outcome
  Reduction of radiofrequency time in the byLAWT arm
Number of application | intraprocedural outcome
  Reduction of the number of application in the byLAWT arm

CONTACTS AND LOCATIONS:
Locations (1):
- Teknon Medical Center, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Teres C, Soto-Iglesias D, Penela D, Jauregui B, Ordonez A, Chauca A, Carreno JM, Scherer C, San Antonio R, Huguet M, Roque A, Ramirez C, Oller G, Jornet A, Palet J, Santana D, Panaro A, Maldonado G, de Leon G, Jimenez G, Evangelista A, Carballo J, Ortiz-Perez JT, Berruezo A. Personalized paroxysmal atrial fibrillation ablation by tailoring ablation index to the left atrial wall thickness: the 'Ablate by-LAW' single-centre study-a pilot study. Europace. 2022 Mar 2;24(3):390-399. doi: 10.1093/europace/euab216. PMID 34480548
- [Result] Duytschaever M, De Pooter J, Demolder A, El Haddad M, Phlips T, Strisciuglio T, Debonnaire P, Wolf M, Vandekerckhove Y, Knecht S, Tavernier R. Long-term impact of catheter ablation on arrhythmia burden in low-risk patients with paroxysmal atrial fibrillation: The CLOSE to CURE study. Heart Rhythm. 2020 Apr;17(4):535-543. doi: 10.1016/j.hrthm.2019.11.004. Epub 2019 Nov 9. PMID 31707159
- [Result] Taghji P, El Haddad M, Phlips T, Wolf M, Knecht S, Vandekerckhove Y, Tavernier R, Nakagawa H, Duytschaever M. Evaluation of a Strategy Aiming to Enclose the Pulmonary Veins With Contiguous and Optimized Radiofrequency Lesions in Paroxysmal Atrial Fibrillation: A Pilot Study. JACC Clin Electrophysiol. 2018 Jan;4(1):99-108. doi: 10.1016/j.jacep.2017.06.023. Epub 2017 Sep 27. PMID 29600792
- [Result] Hussein A, Das M, Riva S, Morgan M, Ronayne C, Sahni A, Shaw M, Todd D, Hall M, Modi S, Natale A, Dello Russo A, Snowdon R, Gupta D. Use of Ablation Index-Guided Ablation Results in High Rates of Durable Pulmonary Vein Isolation and Freedom From Arrhythmia in Persistent Atrial Fibrillation Patients: The PRAISE Study Results. Circ Arrhythm Electrophysiol. 2018 Sep;11(9):e006576. doi: 10.1161/CIRCEP.118.006576. PMID 30354288
- [Derived] Falasconi G, Penela D, Soto-Iglesias D, Latini AC, Landra F, Curti E, Francia P, Saglietto A, Turturiello D, Viveros D, Bellido A, Alderete J, Zaraket F, Franco-Ocana P, Valcher S, Amata F, Valeriano C, Gigante C, Teresi L, Tonello B, Mea R, Sanchez-Molla L, De Lucia C, Huguet M, Camara O, Ortiz-Perez JT, Marti-Almor J, Berruezo A. Personalized pulmonary vein isolation guided by left atrial wall thickness for persistent atrial fibrillation ablation: the PeAF-by-LAWT randomized trial. Europace. 2025 Dec 1;27(12):euaf163. doi: 10.1093/europace/euaf163. PMID 40794635
- [Derived] Falasconi G, Penela D, Soto-Iglesias D, Francia P, Teres C, Saglietto A, Jauregui B, Viveros D, Bellido A, Alderete J, Meca-Santamaria J, Franco P, Gaspardone C, San Antonio R, Huguet M, Camara O, Ortiz-Perez JT, Marti-Almor J, Berruezo A. Personalized pulmonary vein antrum isolation guided by left atrial wall thickness for persistent atrial fibrillation. Europace. 2023 May 19;25(5):euad118. doi: 10.1093/europace/euad118. PMID 37125968